CLINICAL TRIAL: NCT04099407
Title: Pirfenidone in Combination With Standard of Care Treatment in Patients With Advanced Liver Fibrosis. Multicenter, Open Trial Focused on Safety, Fibrosis Efficacy Evaluation, and Pharmacokinetic Data.
Brief Title: Pirfenidone and Advanced Liver Fibrosis.
Acronym: PROMETEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Mexicano para el Estudios de las Enfermedades Hepaticas (Other)
Responsible Party: Principal Investigator, Jorge L Poo, Principal Investigador, Head of Liver Clinic, Grupo Mexicano para el Estudios de las Enfermedades Hepaticas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMETEO Study
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Liver Fibrosis; Chronic Liver Disease
Keywords: Liver fibrosis; Fibrosis treatment; Fibrosis reversibility; Pirfenidone
MeSH Terms: conditions — Liver Cirrhosis | interventions — pirfenidone; Standard of Care

STUDY DESIGN:
Intervention Model Description: This will be a real-life, multicenter, open-label, proof of concept trial to determine the safety and efficacy of 12 months of treatment with PR-PFD in combination with standard of care treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antifibrotic plus standard of care treatment (Experimental): Prolonged release pirfenidone formulation in combination with standard of care treatment.
  Interventions: Drug: Pirfenidone; Other: Standard of care

INTERVENTIONS:
Drug: Pirfenidone — Treatment consist of 600 mg tablets of a prolonged-released formulation of Pirfenidone. Patients are instructed to take medication orally, every 12 h, after breakfast and dinner.
Other: Standard of care — All participants will require to adhere to a standard of care including nutritional support, quarterly medical evaluation to review lab results and adjust medications, bi-annual Fibrotest, FibroScan and liver ultrasound, and annual upper-gastrointestinal endoscopy.

SUMMARY:
Pirfenidone (PFD), an oral antifibrotic drug with anti-inflammatory and anti-oxidant properties, has been granted marketing authorization by the European Medicine Agency and FDA, for the treatment of idiopathic pulmonary fibrosis (IPF). However, few studies have focused on its clinical utilization in patients with advanced hepatic fibrosis. Therefore, Investigators aim to evaluate a prolonged-release PFD formulation (PR-PFD) plus standard of care management on disease progression in patients with advanced liver fibrosis (ALF).

Methods: Patients with diverse chronic liver disease etiology (alcohol-related, hepatitis B or C, autoimmune or fatty liver disease) will be screened with two non invasive liver fibrosis methods (Fibroscan®) and Fibro Test®) and those with ALF (F3 or F4) will be treated for at least 12 months with PR-PFD. Antifibrotic effects Will be assessed at 6 and 12 months; variations greater than 30% in estimated fibrosis scores or 1 point on the METAVIR scale will be considered clinically significant. PFD plasma levels, serum endothelin-1, IL6, TNFα and TGFβ1, Quality of life and fatigue scales will be evaluated. Parametric and non parametric statistics will be utilized and p values lower tan 5% will be considered clinically significant.

DETAILED DESCRIPTION:
The study will be conducted in compliance with International Standard good clinical practices (GCPs) and the Declaration of Helsinki. The protocol was approved by local Institutional Review Board and registered in clinical trials.gov.

Clinical and Laboratory Evaluation Blood counts and liver function tests (bilirubin, albumin, prothrombin time expressed as international normalized ratio (INR), serum transaminases, glucose, and creatinine) are measured at 12-week intervals. Patient's somatometric measurements (height and body weight), vital signs, and frequency of adverse events (AE) are recorded. Liver enzymes will be scored as stable, improving, or worsening.

Study End Points The primary efficacy endpoint is a reduction of fibrosis score by at least 30% either in Fibro Test units or kilo Pascals (kPa) according to hepatic elastography or a reduction of 1 point on the METAVIR scale. Secondary efficacy endpoints include improvement in alanine aminotranferase (ALT) and/or aspartate aminotransferase (AST), albumin, serum concentrations of TGFbeta, IL-1 and IL-6 and endothelin, and Child-Pugh and MELD scores. Worsening MELD is defined as switching from a lower-score to a higher-score and improving as switching from a higher-score to a lower-score, where Group 1 was MELD ≤ 9, Group 2 10-19, and Group 3 > 20.

Primary safety endpoints include clinical side effects, blood profile abnormalities, overall survival, and pharmacokinetic (PK) findings. Secondary safety endpoints included quality of life scores.

Evaluation and Classification of Fibrosis Outcomes Fibrosis-regression profile (FRP): decreases >30% in FT score or 30% in kPa in liver stiffness measurement (LSM) or decreasing 1 point on the METAVIR score comparing baseline and M12 measurements.

Fibrosis-stabilization profile (FSP): stable FT results or kPa measurements (variations lower than 30%) or METAVIR score.

Fibrosis-progression profile (FPP): increases greater than 30% in FT score or kPa or increasing 1 point on METAVIR.

Specific Evaluation and Classification of Biochemical Outcomes Biochemical markers: Blood parameters determined after overnight fasting include: albumin, prothrombin time, total bilirubin, ALT, AST, Alkaline phosphatase (AP), and gamma-glutamyltransferase (GGT), measured in fresh serum within 8h of collection on an automated biochemistry analyzer (Hitachi 917; Roche Diagnostics).

alpha-2-macroglobulin (A2M), apolipoprotein-A1, and haptoglobin levels will be assayed by nephelometry (Image; Beckman Coulter).

Fibro Test®: blinded Fibrotest measurements will be performed on fresh serum and according to the recommended pre-analytic and analytic methods.

Hepatic elastography: Transient Elastography (TE) is performed according to published recommendations using the Fibro-Scan® M probe. LSM is expressed in kPa. Only procedures with at least 10 validated measurements, >60% success rate, and an interquartile range <30% of the median will be considered reliable. Patients with ascites will be offered real time shear wave elastography (Aixplorer, Supersonic Imagine).

Cytokines and pirfenidone: Serum concentrations of Interleukin 6 (IL-6), transforming growth factor beta (TGF-β1), endothelin 1 (ET-1), and tumor necrosis factor alpha (TNF-α) will be quantified by ELISA in an automated enzyme-linked immunosorbent assay (EIA) analyzer Coda Microplate System (Bio-Rad Laboratories, Inc., Hercules, California, USA) and values normalized against serum of healthy volunteers with normal liver function and LSM <5 kPa (F0).

Evaluation of Safety Profile Monitoring for safety and toxicity will be performed throughout the study. When necessary, appropriate medical intervention will be provided.

Quality of life assessment: All patients will fill out the Euro-Qol Index survey, including the visual analog scale evaluation at baseline and at 12 months. Investigators incorporate the nonutility-based Short Form-36v2 survey, which provides a detailed profile of health-related quality of life.

Ethical considerations. The study will be conducted in accordance with the Declaration of Helsinki and the E6 Good Clinical Practice Standards International Conference on Harmonization (ICH).

Statistical Data Analysis: Investigators will be using the Statistical Package for the Social Sciences (SPSS) Statistical software 6.12 for Windows. Descriptive statistics include mean, standard deviation standard error. A paired or unpaired t Test will be used to compare means before and after study medication administration. Values <5% will be considered significant. Kaplan Meier survival analyses will include all patients on active study-medication treatment despite duration of exposure. Sample size calculation was based on the following assumptions: (1) mean expected baseline elastography score of 27.4 kPa, standard deviation of 15.7; expected estimated-fibrosis reduction rate higher than 30% (delta); (4) alpha error of 1%; (5) an accepted beta error of 10% (power = 90%); (6) two tails. The final number of patients required to find a significant difference using the G power statistical program was 61 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic liver disease whose fibrosis continued to progress despite abstaining from alcohol (ALD), achieving sustained virologic response (VHC), or otherwise maintaining stable disease (NAFLD, AIH)..
2. Advanced liver fibrosis defined as fibrosis grade 3 or grade 4 according to METAVIR scale based in two non-invasive liver fibrosis evaluation methods (FibroScan and Fibrotest).
3. Stable liver disease.

Exclusion Criteria:

1. Patients with mild fibrosis (F1-F2)
2. Under medication with colchicine, silymarin, non-steroidal anti-inflammatory drugs, and any hepatotoxic drug.
3. Decompensation based on a history of hepatic encephalopathy, esophageal variceal bleeding, or ascites in the previous 6 months
4. HIV, Hepatitis B virus (HBV) or any active infectious processes not of a self-limited nature.
5. Concomitant or prior history of malignancy other than curatively-treated skin cancer or surgically-cured in situ carcinoma of the cervix.
6. Hemoglobinopathy or any disease associated with hemolysis.
7. History of significant cardiac or pulmonary disease that could be exacerbated by anemia.
8. Liver masses detected by baseline scanner or Alpha-fetoprotein >100 ng/L.
9. Pregnancy.
10. Alcohol or intravenous drug abuse within the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Fibrosis reversal based on Fibrotest | 12 months
  Reduction of fibrosis score by at least 30% in Fibrotest units.
Fibrosis reversal based on Hepatic Elastography | 12 months
  Reduction of fibrosis score by at least 30% in kilo Pascals (kPa) according to accurate hepatic elastography measurements.
Fibrosis reversal based on METAVIR | 12 months
  Reduction of fibrosis score by at least one point on the METAVIR fibrosis scale.
Safety endpoint based on clinical side effects | 12 months
  Clinical side effects wiil be evaluated according to World Health Organization grade modified toxicity scale.

SECONDARY OUTCOMES:
Improvement in Quality of life | 12 months
  Quality of life will be evaluated according to nonutility-based Short Form-36 survey.
Improvement in Liver function values: bilirubin | 12 months
  Improvement by at least 30% in serum Bilirubin levels (mg/dL)
Improvement in Liver function values:albumin | 12 months
  Improvement by at least 30% in serum albumin levels (mg/dL)
Improvement in fibrosis molecular marker | 12 months
  Improvement in serum concentrations of transforming growth factor beta (TGF-β1), quantified by ELISA in an automated enzyme-linked immunosorbent assay (EIA) analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Clinic 1, Mexico City, Mexico

REFERENCES:
- [Derived] Poo JL, Torre A, Aguilar-Ramirez JR, Cruz M, Mejia-Cuan L, Cerda E, Velazquez A, Patino A, Ramirez-Castillo C, Cisneros L, Bosques-Padilla F, Hernandez L, Gasca F, Flores-Murrieta F, Trevino S, Tapia G, Armendariz-Borunda J, Munoz-Espinosa LE. Benefits of prolonged-release pirfenidone plus standard of care treatment in patients with advanced liver fibrosis: PROMETEO study. Hepatol Int. 2020 Sep;14(5):817-827. doi: 10.1007/s12072-020-10069-3. Epub 2020 Aug 19. PMID 32813194